CLINICAL TRIAL: NCT01235468
Title: Allogenic Transplantation of Ex-vivo Expanded CB Progenitors for Haematological Disorders
Brief Title: Allogenic Transplantation of Ex-vivo Expanded Cord Blood (CB)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: loss of support
Sponsor: Dr. Avichai Shimoni MD (Other Government)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor-Investigator, Dr. Avichai Shimoni MD, Dr. Avichai Shimoni, hematologist, Sheba Medical Center
Organization: Sheba Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHEBA-10-7959-AN-CTIL
Record Dates: First submitted 2010-11-02; First posted 2010-11-05 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Umbilical Cord Blood; Stem Cell Transplantation; Hematological Malignancies
Keywords: umbilical cord blood; ex vivo expansion; engraftment; GVHD
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CB expnasion (Experimental): ex-vivo expansion of cord blood for transplantation
  Interventions: Biological: ex vivo expansion

INTERVENTIONS:
Biological: ex vivo expansion — ex-vivo expansion of cord blood for transplantation

SUMMARY:
The aim of this study is to evaluate the safety profile and tolerability of infusion of cord blood cells expanded in the lab and to evaluated whether through the infusion of expanded cells it is possible to expedite engraftment time after transplantation.

DETAILED DESCRIPTION:
Stem cell transplantation is a curative approach for patients with hematological malignancies. Umbilical cord blood is a source of stem cells for transplantation in patients with no related donor. However, in adults, the number of stem cells in a single unit, may be too low to allow engraftment, and the time to engraftment may be prolonged, increasing the risks of the transplant. In this study, we expand part of the cord blood unit, in the lab, trying to increase unit size, such that it would be suitable for adults, and would allow safe engraftment.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* hematological malignancy
* standard indication for allogeneic transplantation
* expected survival time over 12 weeks
* no related or unrelated donor
* availability of a cord blood unit of compatible placental blood cryopreserved in at least 2 different bags; one of the two units should have a cellular content at least equal to the minimum dose of 2 x 107 nucleated cells per kilogram of body weight

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status >2
* Prior allogeneic transplantation
* Pregnant or nursing women
* Positive serology for hepatitis B or C
* HIV positive
* Left ventricular ejection fraction < 50%
* DLCO < 50%
* Psychiatric, addictive, or any disorder/disease which compromises ability to give informed consent for participation in this study
* Treatment with other investigational drugs within 4 weeks of enrolling in this protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Safety | 1 month
  Number of patients with adverse events during infusion
engraftment | 3 months
  Time to engraftment
treatment-related toxicity | 3 months
  Type and severity of adverse events after transplantation using the NCI CTC scale
GVHD | 1 year
  Number of patients with acute and chronic GVHD after transplantation

SECONDARY OUTCOMES:
Immunological reconstruction | 5 years
  immunological reconstruction after transplantation measured by lymphocyte number and function
relapse | 5 years
  rate of disease recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Nagler, MD, Principal Investigator — Chaim Sheba Medical Center